CLINICAL TRIAL: NCT05052671
Title: Application of ctDNA Assay in the Neoadjuvant and Adjuvant Chemotherapy Setting in Patients With Resectable Pancreatic Cancer
Brief Title: ctDNA Assay in Patients With Resectable Pancreatic Cancer
Acronym: OU-SCC-ctDNA
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-ctDNA
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue from core biopsy and blood sample for ctDNA assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the proportion of positive ctDNA -freely circulating tumor DNA fragments found in the blood plasma- in patients with pancreatic cancer and to better understand the relationship between possible ctDNA biomarkers and patient survival. A successful study may provide preliminary evidence that helps improve future patient care through targeted diagnostics, prognosis, and/or treatment.

DETAILED DESCRIPTION:
The objective of this study is to assess the role of serial ctDNA analysis as integrative biomarker in patients with resectable or borderline resectable pancreatic cancer undergoing treatment with curative intent. This is a single arm prospective tissue/blood collection from patients undergoing neoadjuvant treatment and Surgery as well as surveillance, plan to accrue up to 50 patients. Primary objective is to determine the proportion of ctDNA positive in patients with resectable pancreatic cancer and to evaluate the progression free survival (PFS) in subjects with ctDNA positive versus ctDNA negative.

Patients who consent to the study will participate in pre-study exams and tests to find out if they can take part in the study. This includes, but is not limited to, a doctor's visit with medical history and physical evaluation, blood work, pregnancy test for those capable of becoming pregnant, and imaging tests.

The study itself will include the patient's regular treatment for pancreatic cancer which may include 4 to 6 months of chemotherapy, chemo-radiation, surgery to remove pancreatic cancer, 24 weeks of post operative ctDNA surveillance and follow up for 2 years. Blood will be drawn at regular time points during this study for ctDNA detection. The tumor tissue at diagnosis will be collected to develop a personalized and tumor informed PCR test.

ELIGIBILITY:
Inclusion Criteria

1. Newly diagnosed exocrine pancreatic cancer with either pathology or radiology imaging suggestive of adenocarcinoma
2. Resectable/Borderline Resectable Pancreatic cancer as defined by the NCCN guidelines
3. ≥ 18 years old at the time of informed consent
4. ECOG Performance Status 0 or 1
5. Patients who are candidates for neoadjuvant chemo/chemoradiotherapy or upfront surgery are eligible for the study.
6. Ability to provide written informed consent and HIPAA authorization
7. Patients must have a life expectancy of at least 6 months

Exclusion Criteria

1. Patients with pancreatic malignant tumor histologically confirmed as neuroendocrine or any other type of malignancies
2. Positive pregnancy test, pregnant, or breastfeeding
3. Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study
4. Locally advanced or metastatic disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 or over with newly diagnosed exocrine pancreatic cancer with pathology confirmed adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ctDNA Positivity in Patients with Resectable Pancreatic Cancer | Baseline
  Determine the proportion of ct DNA positivity in patients with resectable pancreatic cancer.
Progression free survival (PFS) | 2 years
  Determine PFS in ctDNA positive versus ctDNA negative patients.

SECONDARY OUTCOMES:
Conversion time from ctDNA negative to positive after surgical resection. | 2 years
  Median time from positive ctDNA to negative ctDNA in patients with pancreatic cancer undergoing surgical resection and adjuvant chemotherapy
Median time for select genes to convert from positive to negative. | 2 years
  Median time from any positive KRAS, CDKN2A, SMAD4, or TP53 genes to become negative
Overall survival (OS) in ctDNA positive versus ctDNA negative. | 2 years
  Comparison of overall survival rate of ctDNA positive versus ctDNA negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sagila George, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Stephenson Cancer Center- Tulsa, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No